CLINICAL TRIAL: NCT05407285
Title: A Triple-blind, Placebo-controlled, Randomized, Crossover Study of Low Dose Oral Synthetic Cannabidiol Effects in Healthy Cannabis Occasional Users
Brief Title: A Study of Ingested Cannabidiol in Healthy Occasional Cannabis Users
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22.049
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Crossover Assignment In this crossover design, participants will be administered both dosages of CBD and placebo during participation in the study. Participant will be randomly assigned to one of ten pre-determined sequences with a CBD or placebo product at 5 dosages (0 mg, 20 mg, 50 mg, 100 mg and 200 mg). Participants will be randomized based on a completely balanced 5 by 5 latin square.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0 mg CBD, ingested placebo (Experimental): Ingested placebo containing 0 mg CBD. Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit. The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: cannabis 0 mg, placebo; Drug: Cannabis 20 mg,; Drug: Cannabis 50 mg; Drug: Cannabis 100 mg; Drug: Cannabis 200 mg
- 20 mg CBD, ingested CBD (Experimental): Ingested cannabis containing 20 mg CBD. Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit. The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: cannabis 0 mg, placebo; Drug: Cannabis 20 mg,; Drug: Cannabis 50 mg; Drug: Cannabis 100 mg; Drug: Cannabis 200 mg
- 50 mg CBD, ingested CBD (Experimental): Ingested cannabis containing 50 mg CBD. Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit. The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: cannabis 0 mg, placebo; Drug: Cannabis 20 mg,; Drug: Cannabis 50 mg; Drug: Cannabis 100 mg; Drug: Cannabis 200 mg
- 100 mg CBD, ingested CBD (Experimental): Ingested cannabis containing 100 mg CBD. Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit. The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: cannabis 0 mg, placebo; Drug: Cannabis 20 mg,; Drug: Cannabis 50 mg; Drug: Cannabis 100 mg; Drug: Cannabis 200 mg
- 200 mg CBD, ingested CBD (Experimental): Ingested cannabis containing 200 mg CBD Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit. The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: cannabis 0 mg, placebo; Drug: Cannabis 20 mg,; Drug: Cannabis 50 mg; Drug: Cannabis 100 mg; Drug: Cannabis 200 mg

INTERVENTIONS:
Drug: cannabis 0 mg, placebo — Eligible participant will be randomize 1:1:1:1:1 to receive study products in a prefilled single syringe with 2 ml of product solution with varying amounts of CBD (0 - 20 mg - 50 mg -100 mg - 200 mg. Only one research product will be ingested at each visit. The sequence will depend on the assigned randomization group.
  Other Names: CBD, placebo
Drug: Cannabis 20 mg, — Eligible participant will be randomize 1:1:1:1:1 to receive study products in a prefilled single syringe with 2 ml of product solution with varying amounts of CBD (0 - 20 mg - 50 mg -100 mg - 200 mg. Only one research product will be ingested at each visit. The sequence will depend on the assigned randomization group.
  Other Names: CBD
Drug: Cannabis 50 mg — Eligible participant will be randomize 1:1:1:1:1 to receive study products in a prefilled single syringe with 2 ml of product solution with varying amounts of CBD (0 - 20 mg - 50 mg -100 mg - 200 mg. Only one research product will be ingested at each visit. The sequence will depend on the assigned randomization group.
  Other Names: CBD
Drug: Cannabis 100 mg — Eligible participant will be randomize 1:1:1:1:1 to receive study products in a prefilled single syringe with 2 ml of product solution with varying amounts of CBD (0 - 20 mg - 50 mg -100 mg - 200 mg. Only one research product will be ingested at each visit. The sequence will depend on the assigned randomization group.
  Other Names: CBD
Drug: Cannabis 200 mg — Eligible participant will be randomize 1:1:1:1:1 to receive study products in a prefilled single syringe with 2 ml of product solution with varying amounts of CBD (0 - 20 mg - 50 mg -100 mg - 200 mg. Only one research product will be ingested at each visit. The sequence will depend on the assigned randomization group.
  Other Names: CBD

SUMMARY:
The purposes of this study are 1) to determine if the administration of different low doses of oral CBD (20 mg, 50 mg, 100 mg and 200 mg) result in detectable subjective pleasant drug effect compared to placebo and 2) to qualitatively explore whether low dose of oral CBD is associated with effects that are not detected with the available research tools.

DETAILED DESCRIPTION:
Cannabis contains over 100 cannabinoids, the two most prominent being Δ-9-tetrahydrocannabinol (THC) and cannabidiol (CBD). A growing body of evidence exists surrounding the effects of both THC and CBD, however, less is known about the specific effects of CBD concentrations alone. Most existing data regarding the effects of CBD come from studies where this compound is administered in high doses in a therapeutic context, and where the subject can be administered either CBD, THC or both together. These contexts are not representative of the current use by many consumers. Indeed, several available products contain CBD at much lower doses. The overall objective of this study is to evaluate the acute behavioral and biological effects of low doses of ingested CBD (between 20-200mg) and placebo in occasional cannabis users. Potential outcomes not detected with usual assessment tools designed to evaluate THC-induced effects will also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Between 21 and 65 years of age, inclusively;
2. Occasional users, having used cannabis three days or less in the 28 days prior to enrollment;
3. Be able to provide a signed informed consent;
4. Willing to comply with study procedures and requirements as per protocol, including to abstain from using other cannabis products or any drugs (except alcohol or nicotine) 7 days prior to study visits;
5. Able to communicate and understand English or French language;
6. For female participants:

   a. Without childbearing potential, defined as: i. postmenopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age); or ii. Documented surgically sterilized (i.e., tubal ligation, hysterectomy, or bilateral oophorectomy); or b. With childbearing potential: i. Must have negative pregnancy test result at screening and at subsequent visits.

ii. AND have no pregnancy plan while on the trial. iii. AND agree to use a medically accepted method of birth control throughout the study.

Exclusion Criteria:

1. Any disabling medical condition, as assessed by medical history, physical exam, vital signs and/or laboratory assessments that, in the opinion of the study physician, precludes safe participation in the study or the ability to provide fully informed consent;
2. Known chronic liver disease or aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >ULN (Upper Limit of Normal) at screening visit;
3. Mean systolic blood pressure >180 mmHg (millimeter of mercury);
4. Resting heart rate over 100 beats per minute (bpm);
5. Current body mass index (BMI) of over 40;
6. Must not have any clinically significant ECG abnormalities at screening visit;
7. Severe psychiatric condition (history of schizophrenia, schizoaffective disorder or bipolar disorder; current acute psychosis, mania or current suicidality based on the Mini International Neuropsychiatric Interview);
8. Any other disabling, unstable or acute mental condition that, in the opinion of the study physician, precludes safe participation in the study or ability to provide fully informed consent;
9. Current substance use disorder (except nicotine) according to Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders ( SCID-V);
10. Currently pregnant, breastfeeding or planning to become pregnant either at screening or while enrolled in the study;
11. Pending legal action or other reason that, in the opinion of the study physician, might prevent study completion;
12. Use of medication within 7 days of experimental sessions; which, in the opinion of the Investigator, may interact with CBD,
13. Participation in clinical trials or undergoing other investigational procedure related to cannabis or cannabinoid administration within 30 days prior to randomization.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Pleasant drug effect | T1 (60 minutes after ingestion)
  Pleasant drug effect will be assessed using a single item, visual analog scale, administered following administration of the study product at each study visit. It is rated on a continuous scale ranging from 0 (not at all) to 100 (extremely).
Pleasant drug effect | T2 (120 minutes after ingestion)
  Pleasant drug effect will be assessed using a single item, visual analog scale, administered following administration of the study product at each study visit. It is rated on a continuous scale ranging from 0 (not at all) to 100 (extremely).
Pleasant drug effect | T3 (210 minutes after ingestion)
  Pleasant drug effect will be assessed using a single item, visual analog scale, administered following administration of the study product at each study visit. It is rated on a continuous scale ranging from 0 (not at all) to 100 (extremely).
Pleasant drug effect | T4 (300 minutes after ingestion)
  Pleasant drug effect will be assessed using a single item, visual analog scale, administered following administration of the study product at each study visit. It is rated on a continuous scale ranging from 0 (not at all) to 100 (extremely).
Pleasant drug effect | T5 (360 minutes after ingestion)
  Pleasant drug effect will be assessed using a single item, visual analog scale, administered following administration of the study product at each study visit. It is rated on a continuous scale ranging from 0 (not at all) to 100 (extremely).

SECONDARY OUTCOMES:
Drug Effects associated with cannabis ingestion | T1 (60 minutes after ingestion)
  Drug Effects Questionnaire (twenty-three-item) will be use to assess participant's physical signs, symptoms associated with cannabis ingestion and desire to use cannabis. The Drug Effects Questionnaire uses visual analogue scale, ranging from 0 (not at all) to 100 (extremely).
Drug Effects associated with cannabis ingestion | T2 (120 minutes after ingestion)
  Drug Effects Questionnaire (twenty-three-item) will be use to assess participant's physical signs, symptoms associated with cannabis ingestion and desire to use cannabis. The Drug Effects Questionnaire uses visual analogue scale, ranging from 0 (not at all) to 100 (extremely).
Drug Effects associated with cannabis ingestion | T3 (210 minutes after ingestion)
  Drug Effects Questionnaire (twenty-three-item) will be use to assess participant's physical signs, symptoms associated with cannabis ingestion and desire to use cannabis. The Drug Effects Questionnaire uses visual analogue scale, ranging from 0 (not at all) to 100 (extremely).
Drug Effects associated with cannabis ingestion | T4 (300 minutes after ingestion)
  Drug Effects Questionnaire (twenty-three-item) will be use to assess participant's physical signs, symptoms associated with cannabis ingestion and desire to use cannabis. The Drug Effects Questionnaire uses visual analogue scale, ranging from 0 (not at all) to 100 (extremely).
Drug Effects associated with cannabis ingestion | T5 (360 minutes after ingestion)
  Drug Effects Questionnaire (twenty-three-item) will be use to assess participant's physical signs, symptoms associated with cannabis ingestion and desire to use cannabis. The Drug Effects Questionnaire uses visual analogue scale, ranging from 0 (not at all) to 100 (extremely).
Change in dissociation | Baseline and after ingestion at (120 minutes, 300 minutes)
  Dissociation will be assessed using the Clinician Administered Dissociative States Scale administered at Baseline (T0) and following administration of the study product (T2- 120 minutes, T4-300 minutes) at each study visit. The Clinician Administered Dissociative States Scale, a 28-items validated instrument, includes 5 observer items and 23 participant self-report items rated on a 5-point scale, ranging from 0 (not at all) to 4 (extremely). Minimum score :0 not at all; Maximum score 92 extremely dissociate
Cannabis-Specific Subjective Effects | T5 (360 minutes after ingestion)
  Subjective effects of cannabis will be assessed using both the positive and negative subscales of the Cannabis Experience Questionnaire administered following administration study product. Each item is rated on a 5-point scale, ranging from 1 (not at all) to 5 (severely).The positive subscale includes16 items related to euphoric experiences (maximum 90 and minimum 16). The negative subscale includes 25 items related to paranoid-dysphoric experiences (Maximum 125 and minimum 25).
Change in Affect | Baseline and after ingestion at (120 minutes, 300 minutes)
  Affect will be measured using the Positive and Negative Affect Schedule administered at Baseline (T0) and following administration of the study product at each study visit. The Positive and Negative Affect Schedule is a 20-item validated questionnaire divided into subscales of positive (10 items) and negative affect (10 items). Each item is rated on a 5-point scale ranging from 1 (not at all) to 5 (extremely). For each subscale minimum is 10 and maximum 50.
Change in Anxiety Symptoms | Baseline and after ingestion at (120 minutes, 300 minutes)
  Symptoms of anxiety will be assessed using the States-Trait-Anxiety-Inventory, a 20-item validated self-report scale that measures the severity of anxiety in adults. Each symptom is rated on a 4-point scale ranging from 1 (not at all) to 4 (very much).
Change in the incidence of Treatment Emergent-adverse Events | Baseline and after ingestion at (60 minutes, 120 minutes, 210 minutes, 300 minutes, 360 minutes)
  Adverse events will be collected prior to administration of the study product (T0) and following administration of the study product (T1, T2, T3,T4, T5)
Change on cognition | Baseline and after ingestion at 210 minutes
  The Cambridge Neuropsychological Test Automated Battery tests will be used for the rapid assessment of multiple cognitive components.
Visit Intoxication Assessment | End of the visit, approximatively 360 minutes after ingestion
  Signs of intoxication will be assess using the modified Standardized Field Sobriety Test.

OTHER OUTCOMES:
Change in plasma concentration of CBD | Baseline and after ingestion at ( 60 minutes, 120 minutes, 210 minutes, 300 minutes, 360 minutes)
  Plasma levels of CBD will be determined by high performance liquid chromatography-tandem mass spectrometry at baseline and after ingestion.
Change in plasma concentration of 7-Hydroxy-cannabidiol | Baseline and after ingestion at ( 60 minutes, 120 minutes, 210 minutes, 300 minutes, 360 minutes)
  Plasma levels of CBD will be determined by high performance liquid chromatography-tandem mass spectrometry at baseline and after ingestion.
Change in plasma concentration of 7-Carboxy-Cannabidiol | Baseline and after ingestion at ( 60 minutes, 120 minutes, 210 minutes, 300 minutes, 360 minutes)
  Plasma levels of CBD will be determined by high performance liquid chromatography-tandem mass spectrometry at baseline and after ingestion.
Change in plasma concentration of Anandamide | Baseline and after ingestion at ( 60 minutes, 120 minutes, 210 minutes, 300 minutes, 360 minutes)
  Plasma levels of CBD will be determined by high performance liquid chromatography-tandem mass spectrometry at baseline and after ingestion.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, MD,MS, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre de recherche du Centre Hospitalier Universitaire de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abboud A, Chester LA, Hebert FO, Jutras-Aswad D. Sex-specific association between low oral doses of cannabidiol (CBD) and plasma concentration of anandamide (AEA), N-palmitoylethanolamine (PEA) and N-oleoylethanolamine (OEA) in healthy occasional cannabis users. J Cannabis Res. 2026 Jan 9;8(1):20. doi: 10.1186/s42238-025-00356-x. PMID 41514385